CLINICAL TRIAL: NCT03132077
Title: Retrospective Analysis of Patient Outcome Questionnaire Following Primary Knee Replacement
Brief Title: Analysis of Patient Outcome Questionnaire Following Primary Knee Replacement
Status: Completed | Type: Observational
Sponsor: University of Salford (Other)
Collaborators: Stockport NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Bodor Bin sheeha, Principal Investigator -PhD student at University of Salford, University of Salford
Other Study IDs: usalford- retrospective
Record Dates: First submitted 2017-04-11; First posted 2017-04-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- satisfaction post total knee arthroplasty: The focus of this project is exploring outcomes post-primary total knee arthroplasty (TKA) using the available pre/post-operative Oxford Knee Score (OKS), University of California Los Angeles (UCLA) Activity Score, EQ-5D General Health Questionnaire, Visual Analogue (VAS) for pain, age and smoking status data, and correlations between these data and post operation patient satisfaction.
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — surgical intervention for end stage of knee osteoarthritis
  Other Names: total knee replacement surgery

SUMMARY:
The intention is to explore whether there are factors which help us to understand why some patient outcomes are not successful and identify prediction factors for progression. It will also assess the available outcomes pre- and post-surgery may explore prediction tools for good/poor progression and improve the patient's selection, patient preparation or timing for surgery.

The focus of this project is exploring outcomes post-primary total knee arthroplasty (TKA) using the available pre/post-operative Oxford Knee Score (OKS), University of California Los Angeles (UCLA) Activity Score, EQ-5D General Health Questionnaire, Visual Analogue (VAS) for pain, age and smoking status data, and correlations between these data and post operation patient satisfaction.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a major cause of disability around the world; it is the most common chronic condition in primary care in the UK. By 2030 it is predicted to be the greatest cause of disability in the general population. An effective end-stage treatment for knee OA is knee-replacement surgery.

In England and Wales, the number of knee-replacement procedures recorded by the National Joint Registry in 2013 was 91,703, which represents an increase of 0.9 % over 2012. The data analysis by the National Joint Registry and the Office of National Statistics suggests that, by 2030, primary TKAs will increase by 117% from the 2012 level. Subsequently, TKA revision surgeries are expected to increase incrementally by 332%.

Post-TKA, 75-85% of patients report satisfaction with surgery outcomes, while the remaining 15-25% are dissatisfied. Total knee arthroplasty's success has traditionally been evaluated from the surgeon's perspective, e.g. the presence of surgical complications or implant survival. This is gradually changing to involve the patient in measuring health outcomes and decision-making processes. Patient-reported outcome measures (PROMs) have evolved to explore patient perspectives by monitoring the quality of care in health organizations and conducting clinical trial outcomes. National Health Service used PROMs to measures health gain in patients undergoing hip replacement, knee replacement, varicose vein and groin hernia surgery in England, based on responses to questionnaires before and after surgery.

This retrospective cohort study will investigate outcomes 1 and 3 years post-TKA, and factors that may predict good/poor progression based on previously gathered data, which may minimize the effect of prospective data collection bias. The study will explore accurate prediction factors of post-TKA satisfaction at Stockport NHS Foundation Trust operates at Stepping Hill Hospital which is a busy District General Hospital, with a large orthopaedic department. Outcome following knee replacement surgery is closely monitored and matches the best performing units in the UK. Potentially, reliable outcome prediction could, however, improve patient selection for surgery, as appropriate timing for surgery depends on patient symptoms and efficient patient preparation for surgery if it is to be cost-effective. Accurate preoperative prediction is crucial to minimize the potential for unrealistic expectations which may improve their satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* The present study is a retrospective randomised analysis of outcomes 1 years post-TKA.
* All individuals have previously consented to give access to their data for research studies.
* All patients' records prospectively gathered data spanning more than 3 years will be reviewed, if they were scheduled for primary unilateral TKA for end-stage knee osteoarthritis and were in a stable and controlled medical condition at Stepping Hill Hospital.
* The records will be considered eligible if the following criteria are met:

  * At least one preoperative record no more than 6 months prior to the surgery, 1-year postoperative records available.
  * In regards to the questionnaires, (OKS, UCLA and EQ-5D), a maximum of one missing question for UCLA and two for OKS questionnaire.

Exclusion Criteria:

Potential research records were excluded from the study if;

* The patient had more than acceptable missing datum for any outcome score.
* The patient did not consent to the use of their records for research purposes.
* No preoperative record or the postoperative records not available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The inclusion of a minimum of 400 patient records-comprising both males and females-is planned, to achieve 80% power to detect associations between preoperative factors and post-TKA outcomes at the 5% level and a correlation coefficient of 0.2. This will explore the prediction factors that account for more than 4% of outcome variation, that less than oxford knee score clinically detectable changes (Cohen, 1988).
Sampling Method: Probability Sample
Enrollment: 1301 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in Patient's Report Outcome Measures (Oxford knee score) before and after the surgery | 1-3 years post total knee arthroplasty
  To explore factors which may help us understand why some patient outcomes are not successful and identify factors associated with poor satisfaction using Oxford knee score (OKS) as patients report outcome measures at Stepping Hill Hospital, Stockport

SECONDARY OUTCOMES:
Changes in Patient's Report Outcome Measures- University of California Los Angeles (UCLA) activity score- before and after the surgery | 1-3 years post total knee arthroplasty
  To explore factors which may help us understand why some patient outcomes are not successful and identify factors associated with poor satisfaction using University of California Los Angeles (UCLA) activity score as patients report outcome measures at Stepping Hill Hospital, Stockport
Changes in Patient's Report Outcome Measures -EQ-5D general health questionnaire - before and after the surgery | 1-3 years post total knee arthroplasty
  To explore factors which may help us understand why some patient outcomes are not successful and identify factors associated with poor satisfaction using EQ-5D general health questionnaire as patients report outcome measures at Stepping Hill Hospital, Stockport
Changes in Patient's Report Outcome Measures - visual analogue scales (VAS) - before and after the surgery | 1-3 years post total knee arthroplasty
  To explore factors which may help us understand why some patient outcomes are not successful and identify factors associated with poor satisfaction using visual analogue scales (VAS) as patients report outcome measures at Stepping Hill Hospital, Stockport

CONTACTS AND LOCATIONS:
Locations (1):
- Stockport NHS Foundation Trust, Stockport, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bade MJ, Wolfe P, Zeni JA, Stevens-Lapsley JE, Snyder-Mackler L. Predicting poor physical performance after total knee arthroplasty. J Orthop Res. 2012 Nov;30(11):1805-10. doi: 10.1002/jor.22140. Epub 2012 Apr 26. PMID 22539338
- [Background] Brown K, Kachelman J, Topp R, Quesada PM, Nyland J, Malkani A, Swank AM. Predictors of functional task performance among patients scheduled for total knee arthroplasty. J Strength Cond Res. 2009 Mar;23(2):436-43. doi: 10.1519/JSC.0b013e318198fc13. PMID 19197199
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Cohen, J. (1988). Statistical Power Analysis for the Behavioral Sciences USA: LAWRENCE ERLBAUM ASSOCIATES.
- [Background] Field, A. (2009). Discovering Statistics Using SPSS: SAGE Publications Ltd,.
- [Background] Hossain FS, Konan S, Patel S, Rodriguez-Merchan EC, Haddad FS. The assessment of outcome after total knee arthroplasty: are we there yet? Bone Joint J. 2015 Jan;97-B(1):3-9. doi: 10.1302/0301-620X.97B1.34434. PMID 25568406
- [Background] Jagger, C., Matthews, R., Spiers, N., Brayne, C., Comas - Herrera, A., Robinson, T., . . . Croft, P. (2006). Compression or expansion of disability?: forecasting future disability levels under changing patterns of diseases: King's Fund.
- [Background] Klit J, Jacobsen S, Rosenlund S, Sonne-Holm S, Troelsen A. Total knee arthroplasty in younger patients evaluated by alternative outcome measures. J Arthroplasty. 2014 May;29(5):912-7. doi: 10.1016/j.arth.2013.09.035. Epub 2013 Oct 1. PMID 24269097
- [Background] Lungu E, Desmeules F, Dionne CE, Belzile EL, Vendittoli PA. Prediction of poor outcomes six months following total knee arthroplasty in patients awaiting surgery. BMC Musculoskelet Disord. 2014 Sep 8;15:299. doi: 10.1186/1471-2474-15-299. PMID 25201448
- [Background] Noiseux NO, Callaghan JJ, Clark CR, Zimmerman MB, Sluka KA, Rakel BA. Preoperative predictors of pain following total knee arthroplasty. J Arthroplasty. 2014 Jul;29(7):1383-7. doi: 10.1016/j.arth.2014.01.034. Epub 2014 Feb 7. PMID 24630598
- [Background] Patel A, Pavlou G, Mujica-Mota RE, Toms AD. The epidemiology of revision total knee and hip arthroplasty in England and Wales: a comparative analysis with projections for the United States. A study using the National Joint Registry dataset. Bone Joint J. 2015 Aug;97-B(8):1076-81. doi: 10.1302/0301-620X.97B8.35170. PMID 26224824
- [Background] Portney, L., & Watkins, M. (2009). Foundations of Clinical Research: Applications to Practice. London: Pearson/Prentice Hall, 2009.